CLINICAL TRIAL: NCT03011021
Title: Phase 1/ Phase 2 Study of the Therapeutic Effect of Ex-vivo Expanded Umbilical Cord Blood Regulatory T Cells With Liraglutide on Autoimmune Diabetes
Brief Title: Safety and Efficacy of Umbilical Cord Blood Regulatory T Cells Plus Liraglutide on Autoimmune Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Principal Investigator, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Type1 Diabetes Mellitus; Autoimmune Diabetes
Keywords: Autoimmune Diabetes; Umbilical Cord Blood Regulatory T Lymphocyte; Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide; Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UCB-Treg plus Liraglutide (Experimental): Subjects will receive a single infusion of ex vivo expanded umbilical cord blood derived Treg product (2 x 10^6). Dose escalation of liraglutide up to 1.2 mg will be started 3 days after Treg infusion only if no severe side effects showed. Subjects continue to receive the reached liraglutide dose once daily for 6 months thereafter. Insulin will be continued as a routine therapy.
  Interventions: Drug: Liraglutide; Biological: UCB-Treg; Drug: Insulin
- UCB-Treg (Active Comparator): Subjects will receive a single infusion of ex vivo expanded Treg product (2 x 10^6). Insulin will be continued as a routine therapy.
  Interventions: Biological: UCB-Treg; Drug: Insulin
- Liraglutide (Active Comparator): Patients will be subjected to a dose escalation of liraglutide up to 1.2 mg, then continue to receive the reached liraglutide dose once daily for 6 months thereafter. Insulin will be continued as routine therapy.
  Interventions: Drug: Liraglutide; Drug: Insulin
- Insulin (Active Comparator): Patients will receive insulin injection as a routine therapy.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Liraglutide — Dose escalation of Liraglutide starts from 0.6 mg up to 1.2 mg per day.
  Arms: Liraglutide; UCB-Treg plus Liraglutide
Biological: UCB-Treg — Receive Treg infusion: 1~5*10^6/kg b.w. in 100ml normal saline
  Arms: UCB-Treg; UCB-Treg plus Liraglutide
Drug: Insulin — Receive insulin following clinician's instruction.

SUMMARY:
The purpose of this study is to investigate the safety and therapeutic effect of ex-vivo expanded umbilical cord blood regulatory T cells adjunct with Liraglutide on autoimmune diabetes.

DETAILED DESCRIPTION:
Autoimmune Diabetes Mellitus (AIDM) is a subtype of diabetes mellitus caused by autoimmune destruction of beta cells in the islet, including Type 1 diabetes and Latent Autoimmune Diabetes in Adults (LADA). Insulin has been used as a routine therapy for AIDM to alleviate the hyperglycemic status, yet cannot effectively prevent the progressing destruction of beta cells or preserve its function. Regulatory T cells expanded from umbilical cord blood (UCB-Treg) ex-vivo have shown strong capacity to control immune responses in autoimmune diseases, offering a hopeful therapeutic way for AIDM. Glucagon-like peptide (GLP-1) analog Liraglutide has been tested in large-scale clinical trial to prove its various benefits for beta cells and glucolipid metabolism in Type 2 diabetes and obesity patients. However, its clinical application in AIDM is not well-defined so far. The aim of this study is to investigate the potential use of Liraglutide with UCB-Treg infusion in AIDM and examine the safety and efficacy of this new therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to ADA criteria <3 years.
* Age≥ 18 years.
* Positive for at least one of the anti-islet autoantibodies: GADA, IA2A, ZnT8A
* Fasting or postprandial plasma C-peptide more than 100 pmol/L
* Written informed consent from the patient or family representative.

Exclusion Criteria:

* History or family history of medullary thyroid carcinoma or MEN 2 syndrome;
* History of chronic or acute pancreatitis;
* Allergic to liraglutide or any components in Victoza®;
* Hepatic abnormalities (transaminase > 2 times normal);
* Renal impairments (serum creatinine >133 umol/L);
* Cardiovascular diseases (hypertension, coronary heart disease, etc.);
* Presence of anemia (Hb ≤100g/L), leukopenia (<3.5×109/L);
* Presence of disorder in coagulation or anticoagulation, or thrombocytopenia (platelets <100×109/L);
* Presence of acute metabolic disorders; In the case of acute ketone acidosis, with blood ketone over 0.3mmol/L and pH lower than 7.30;
* Presence of any kind of chronic infection or immune deficiency, including hepatitis B, hepatitis C, HIV, syphilis or tuberculosis, etc.;
* Chronic use of systemic glucocorticoids or other immunosuppressive agents for over 3 months;
* Any history of malignancy;
* Female patients who are pregnant or breastfeeding; any female who is unwilling to use a reliable and effective form of contraception for 2 years after recruitment;
* Presence of any infectious diseases, including active skin infections, flu, fever, upper or lower respiratory tract infections; those who wish to participate in the study should keep the infection under control for at least 1 week before receiving Treg product infusion;
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Adverse effects | 2 years
  Primary outcome measures will be the number of participants with adverse events, laboratory abnormalities and other signs of toxicity. Particular focus will be on the number and severity of infusion reactions, complications related to infection, and any potential negative impact on the course of diabetes.

SECONDARY OUTCOMES:
Change in HbA1C | 2 years
  Measure the HbA1C level after treatment
Change in C-peptide | 2 years
  Measure the C-peptide level after treatment
Change in insulin dose | 2 years
  Measure insulin dose patient used after treatment
Hypoglycaemic events | 2 years
  Measure the number of participants with Hypoglycaemic events
Change in titer of autoantibodies | 2 years
  Measure the titer of antoantibodies of participant after treatment
Change in immune cells diversities and quantities. | 2 years
  Measure the immune cells diversities and quantities after treatment
Change in autoimmune-related cytokines | 2 years
  Measure the change of autoimmune- related cytokines after treatment
Life quality evaluation | 2 years
  Number of participants with disturbance of emotion, sleep, resting or energy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD/PhD, Principal Investigator — Second Xiangya Hospital; Haibo Yu, MD/PhD, Principal Investigator — Second Xiangya Hospital
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Milward K, Issa F, Hester J, Figueroa-Tentori D, Madrigal A, Wood KJ. Multiple unit pooled umbilical cord blood is a viable source of therapeutic regulatory T cells. Transplantation. 2013 Jan 15;95(1):85-93. doi: 10.1097/TP.0b013e31827722ed. PMID 23263503
- [Background] Fan H, Yang J, Hao J, Ren Y, Chen L, Li G, Xie R, Yang Y, Gao F, Liu M. Comparative study of regulatory T cells expanded ex vivo from cord blood and adult peripheral blood. Immunology. 2012 Jun;136(2):218-30. doi: 10.1111/j.1365-2567.2012.03573.x. PMID 22348606
- [Background] Brunstein CG, Miller JS, Cao Q, McKenna DH, Hippen KL, Curtsinger J, Defor T, Levine BL, June CH, Rubinstein P, McGlave PB, Blazar BR, Wagner JE. Infusion of ex vivo expanded T regulatory cells in adults transplanted with umbilical cord blood: safety profile and detection kinetics. Blood. 2011 Jan 20;117(3):1061-70. doi: 10.1182/blood-2010-07-293795. Epub 2010 Oct 15. PMID 20952687
- [Background] Rondas D, D'Hertog W, Overbergh L, Mathieu C. Glucagon-like peptide-1: modulator of beta-cell dysfunction and death. Diabetes Obes Metab. 2013 Sep;15 Suppl 3:185-92. doi: 10.1111/dom.12165. PMID 24003936
- [Background] Chang TJ, Tseng HC, Liu MW, Chang YC, Hsieh ML, Chuang LM. Glucagon-like peptide-1 prevents methylglyoxal-induced apoptosis of beta cells through improving mitochondrial function and suppressing prolonged AMPK activation. Sci Rep. 2016 Mar 21;6:23403. doi: 10.1038/srep23403. PMID 26997114
- [Background] Zoso A, Serafini P, Lanzoni G, Peixoto E, Messinger S, Mantero A, Padilla-Tellez ND, Baidal DA, Alejandro R, Ricordi C, Inverardi L. G-CSF and Exenatide Might Be Associated with Increased Long-Term Survival of Allogeneic Pancreatic Islet Grafts. PLoS One. 2016 Jun 10;11(6):e0157245. doi: 10.1371/journal.pone.0157245. eCollection 2016. PMID 27285580